CLINICAL TRIAL: NCT04825522
Title: The Effect of Intrawound Vancomycin Powder in Spine Surgery: A Prospective Randomized Controlled Trial
Brief Title: The Effect of Intrawound Vancomycin Powder in Spine Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Windsor-Essex Compassionate Care Community (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Soliman, Assistant Professor of Neurosurgery, General Neurosurgery Clinical Fellow, Principle Investigator, Windsor-Essex Compassionate Care Community
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB# 21-393
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Experimental Group: For surgeries involving one level, 500mg of vancomycin will be applied. For surgeries involving greater than 1 level and less than 3 levels, 1gm will be applied and for surgeries greater than 3 levels, 2gms will be applied.
  Control Group: Will not receive any extra treatment.
Who Masked: Participant
Masking Description: The patients will not know if they received vancomycin or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Participants will not be receiving vancomycin.
- Vancomycin (Active Comparator): For surgeries involving one level, 500mg of vancomycin will be applied. For surgeries involving greater than 1 level and less than 3 levels, 1gm will be applied and for surgeries greater than 3 levels, 2gms will be applied.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — During spinal surgery, participants will receive intrawound vancomycin powder in their wound before closure.
  Other Names: Treatment group
  Arms: Vancomycin

SUMMARY:
Problem: Postoperative wound infection following various spinal surgeries is a serious complication. The incidence of post-surgical wounds in spine surgery is high, and various researchers have reported different infection rates. In addition, increased healthcare costs, prolonged lengths of stay in hospital, and reduced quality of life as a result of surgical site infections (SSI) are also major concerns. Several methods for avoiding SSI, such as betadine irrigation, vacuum-assisted closure, and intra-wound vancomycin powder, have been used to reduce the rate of wound infection in spine surgery. Use of local vancomycin has been popular because of its protective effects and lower cost. According to some reports, prophylactic administration of intra-wound vancomycin powder before wound closure is an effective method for decreasing postoperative wound infection rates; however, other studies have revealed a non-significant effect of intra-wound vancomycin use for decreasing the postsurgical wound infection rate.

Solution: Therefore, the investigators will prospectively randomize all various types of spinal surgeries to patients who will receive intrawound vancomycin powder and control group who will not receive the powder and to see it's effect in reducing the post-surgical infection.

DETAILED DESCRIPTION:
Potential participants will be identified at the clinic, emergency department, or on the floor by history, clinical examination, and positive imaging findings. The surgeon will notify the study coordinator of the potential patient. The study coordinator will introduce the trial to the patient and obtain informed consent at the office during the clinic visit or his hospital stay. Patient's pre-operative data such as demographics (age and sex), presence of comorbidities like diabetes, ischemic heart disease, asthma patients on steroids, nutrition status using serum albumin level, and previous posterior spine surgical procedures at the operative level will be collected once the patient admitted prior to the procedure. The study coordinator will enroll the patient into the trial, and provide the appropriate intervention (vancomycin application, or no application) using the closed envelope technique of randomization to the neurosurgeon performing the procedure. Patients will also be blinded to avoid the placebo effect. All patients will receive the standard systemic antibiotic prophylaxis. The duration of the procedure, estimated blood loss, type of the procedure (instrumented versus non-instrumented) and the number of levels will be recorded. After the intervention, wound infections will be monitored during a follow-up period of 12 weeks from the date of surgery. Cultured organisms and subsequent treatments will be recorded. The primary outcome is the incidence of infection (either in-patient or in the follow-up). The secondary outcome is the development of other complications including Vancomycin related.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring surgery due to any spine disease.

Exclusion Criteria:

* A previous history of infections at the spine surgical site.
* Biopsy procedure.
* Patients with a postoperative follow-up time of less than 12 weeks.
* Patients allergic to vancomycin.
* Patient is less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1643 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Infection | 3 months
  Number of patients with post-operative wound infection after spinal surgery (including the type of organism and duration of the procedure). Investigators will prospectively randomize all various types of spinal surgeries to patients who will receive intrawound vancomycin powder and control group who will not receive the powder and to see it's effect in reducing the post-surgical infection.

SECONDARY OUTCOMES:
Complications | 3 months
  Number of patients who developed any complications related to the vancomycin.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Soliman, MD, Principal Investigator — Western University
Locations (2):
- Windsor Regional Hospital - Ouellette, Windsor, Ontario, Canada
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie LL, Zhu J, Yang MS, Yang CY, Luo SH, Xie Y, Pu D. Effect of Intra-wound Vancomycin for Spinal Surgery: A Systematic Review and Meta-analysis. Orthop Surg. 2017 Nov;9(4):350-358. doi: 10.1111/os.12356. PMID 29178308
- [Background] Tomov M, Mitsunaga L, Durbin-Johnson B, Nallur D, Roberto R. Reducing surgical site infection in spinal surgery with betadine irrigation and intrawound vancomycin powder. Spine (Phila Pa 1976). 2015 Apr 1;40(7):491-9. doi: 10.1097/BRS.0000000000000789. PMID 25608241
- [Background] Evaniew N, Khan M, Drew B, Peterson D, Bhandari M, Ghert M. Intrawound vancomycin to prevent infections after spine surgery: a systematic review and meta-analysis. Eur Spine J. 2015 Mar;24(3):533-42. doi: 10.1007/s00586-014-3357-0. Epub 2014 May 18. PMID 24838506
- [Background] Hey HWD, Thiam DW, Koh ZSD, Thambiah JS, Kumar N, Lau LL, Liu KG, Wong HK. Is Intraoperative Local Vancomycin Powder the Answer to Surgical Site Infections in Spine Surgery? Spine (Phila Pa 1976). 2017 Feb 15;42(4):267-274. doi: 10.1097/BRS.0000000000001710. PMID 28207669
- [Background] O'Neill KR, Smith JG, Abtahi AM, Archer KR, Spengler DM, McGirt MJ, Devin CJ. Reduced surgical site infections in patients undergoing posterior spinal stabilization of traumatic injuries using vancomycin powder. Spine J. 2011 Jul;11(7):641-6. doi: 10.1016/j.spinee.2011.04.025. Epub 2011 May 19. PMID 21600853